CLINICAL TRIAL: NCT02653768
Title: STepped Exercise Program for Knee Osteoarthritis (STEP-KOA)
Brief Title: STepped Exercise Program for Knee OsteoArthritis
Acronym: STEP-KOA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IIR 14-091
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2020-04-07 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, Knee; Exercise
MeSH Terms: conditions — Osteoarthritis, Knee; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- STEP-KOA (Experimental): This is a stepped exercise program. It begins with an internet-based exercise training program (STEP 1). After three months, participants are assessed to see if they have achieved clinically meaningful improvement in key osteoarthritis outcomes. If so, they remain at STEP 1. If not, they move on to STEP 2, which adds telephone-based coaching. Participants are assessed again three months later. Those that still have not achieved clinically relevant improvement move on to STEP 3, which adds a series of in-person physical therapy visits.
  Interventions: Behavioral: Stepped Exercise Program
- Arthritis Education (AE) (Active Comparator): Participants in the AE control group will receive low literacy educational materials via mail every two weeks. Because STEP-KOA is a multi-component intervention, with participants receiving different numbers of Steps, it is not possible to implement a control condition that will mirror the exact intervention "dose" received by all participants in the STEP-KOA group. However, AE will achieve the goal of providing an active, OA-related control condition.
  Interventions: Behavioral: Arthritis Education

INTERVENTIONS:
Behavioral: Stepped Exercise Program — STEP 1: Participants have access to an internet-based exercise program for knee OA.
  STEP 2: Participants have access to an internet-based exercise program for knee OA plus telephone support.
  STEP 3: Participants have access to an internet-based exercise program for knee OA plus in-person physical therapy visit
  Other Names: STEP-KOA
  Arms: STEP-KOA
Behavioral: Arthritis Education — The arthritis education intervention will include bi-weekly mailings of low-literacy educational materials on a comprehensive set of topics related to OA and its management, based on established treatment guidelines.
  Other Names: AE
  Arms: Arthritis Education (AE)

SUMMARY:
Knee osteoarthritis (OA) is one of the most common chronic conditions and a leading cause of disability among Veterans. Although exercise is known to improve pain, physical abilities, and other outcomes for patients who have knee OA, most individuals with this condition are physically inactive. Therefore there is a need to develop programs that will help Veterans and others with knee OA to increase activity levels. This study will examine a stepped approach to helping Veterans with knee OA to increase physical activity, with increasing levels of program intensity when needed for individual patients to meaningfully improve pain and physical function.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a leading cause of pain and disability among Veterans, and Department of Veterans Affairs health care users are the most severely affected. There is ample evidence that exercise improves pain, function, and other outcomes among patients with knee OA. However, the vast majority of individuals with knee OA are physically inactive. There is clearly a need to develop and implement programs that efficiently and effectively foster regular physical activity and improve key patient-centered outcomes among Veterans with knee OA. This objective of this study is to evaluate the effectiveness a novel STepped Exercise Program for Knee OsteoArthritis (STEP-KOA).

This will be a randomized controlled trial of n=345 Veterans with symptomatic knee OA in two VA Integrated Networks (VISN) 6 sites, with participants assigned to two study arms: STEP-KOA and Arthritis Education Control (AE). STEP-KOA will begin with three months of access to a low-resource internet-based exercise training program that uses patient-specific information to determine and deliver an appropriate personalized exercise plan (Step 1). Participants who do not meet response criteria for clinically meaningful improvement in pain and function after three months of Step 1 will additionally receive telephone calls from an exercise counselor for three months, to facilitate adherence and address barriers to physical activity (Step 2). Participants who still fail to meet response criteria after Step 2 will receive in-person physical therapy visits, which address specific functional impairments and further tailor exercise recommendations (Step 3). Outcomes will be assessed at baseline, 3-months, 6-months, and 9 months (primary outcome time point). Veterans in the AE group will be offered participation in STEP-KOA after completing study assessments. The primary outcome will be the Western Ontario and McMasters Universities Osteoarthritis Index (WOMAC), a measure of lower extremity pain, stiffness and function. The secondary outcomes will be objective measures of physical function. The main study analyses will compare the STEP-KOA intervention to the AE control condition at follow-up time points. The investigators will also evaluate patient characteristics associated with the need for progression to each Step and will conduct a cost-effectiveness analysis of STEP-KOA. This stepped exercise intervention is matched with patient needs, and it also provides the VA with a potential approach for focusing limited physical therapy resources toward patients who do not respond adequately to initial, less resource intensive and costly strategies to improve physical activity and related outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Veteran enrolled at the Durham VA Medical Center (VAMC)
* Physician diagnosis of knee osteoarthritis
* Current knee joint symptoms

Exclusion Criteria:

* Currently meeting physical activity guidelines
* Currently completing Physical Therapy (PT) visits for knee OA
* Gout (in knee)
* Rheumatoid arthritis, fibromyalgia, or other systemic rheumatic disease
* Dementia
* Psychosis
* Active substance abuse disorder
* Meniscus or anterior cruciate ligament (ACL) tear in the past 6 months
* Total joint replacement, other major lower extremity surgery in the past 6 months or planned in the next 9 months
* Severe hearing impairment
* Serious/terminal illness
* Other health problem that would prohibit participation in the study and/or warrant immediate PT
* Current participation in another OA intervention study
* Unstable angina
* History of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (two hospitalizations within the previous 12 months and/or on oxygen)
* Uncontrolled hypertension (diastolic blood pressure >110 mm/Hg or systolic > 200mm/Hg)
* Stroke with moderate to severe aphasia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-07-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli Dominick Allen, PhD, Principal Investigator — Durham VA Medical Center, Durham, NC
Locations (1):
- Durham VA Medical Center, Durham, NC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Allen KD, Bongiorni D, Caves K, Coffman CJ, Floegel TA, Greysen HM, Hall KS, Heiderscheit B, Hoenig HM, Huffman KM, Morey MC, Ramasunder S, Severson H, Smith B, Van Houtven C, Woolson S. STepped exercise program for patients with knee OsteoArthritis (STEP-KOA): protocol for a randomized controlled trial. BMC Musculoskelet Disord. 2019 May 28;20(1):254. doi: 10.1186/s12891-019-2627-8. PMID 31138256
- [Result] Boucher NA, Zullig LL, Shepherd-Banigan M, Decosimo KP, Dadolf J, Choate A, Mahanna EP, Sperber NR, Wang V, Allen KA, Hastings SN, Van Houtven CH. Replicating an effective VA program to train and support family caregivers: a hybrid type III effectiveness-implementation design. BMC Health Serv Res. 2021 May 6;21(1):430. doi: 10.1186/s12913-021-06448-7. PMID 33952263
- [Result] Hughes JM, Bartle JT, Choate AL, Mahanna EP, Meyer CL, Tucker MC, Wang V, Allen KD, Van Houtven CH, Hastings SN. Walking All over COVID-19: The Rapid Development of STRIDE in Your Room, an Innovative Approach to Enhance a Hospital-Based Walking Program during the Pandemic. Geriatrics (Basel). 2021 Nov 10;6(4):109. doi: 10.3390/geriatrics6040109. PMID 34842733
- [Result] Beauchamp T, Arbeeva L, Cleveland RJ, Golightly YM, Hales DP, Hu DG, Allen KD. Accelerometer-Based Physical Activity Patterns and Associations With Outcomes Among Individuals With Osteoarthritis. J Clin Rheumatol. 2022 Mar 1;28(2):e415-e421. doi: 10.1097/RHU.0000000000001750. PMID 33902099
- [Result] Allen KD, Woolson S, Hoenig HM, Bongiorni D, Byrd J, Caves K, Hall KS, Heiderscheit B, Hodges NJ, Huffman KM, Morey MC, Ramasunder S, Severson H, Van Houtven C, Abbate LM, Coffman CJ. Stepped Exercise Program for Patients With Knee Osteoarthritis : A Randomized Controlled Trial. Ann Intern Med. 2021 Mar;174(3):298-307. doi: 10.7326/M20-4447. Epub 2020 Dec 29. PMID 33370174
- [Result] Kaufman BG, Allen KD, Coffman CJ, Woolson S, Caves K, Hall K, Hoenig HM, Huffman KM, Morey MC, Hodges NJ, Ramasunder S, van Houtven CH. Cost and Quality of Life Outcomes of the STepped Exercise Program for Patients With Knee OsteoArthritis Trial. Value Health. 2022 Apr;25(4):614-621. doi: 10.1016/j.jval.2021.09.018. Epub 2021 Oct 29. PMID 35365305

RESULTS

PARTICIPANT FLOW:
Groups:
- STEP-KOA: This is a stepped exercise program. It begins with an internet-based exercise training program (STEP 1). After three months, participants are assessed to see if they have achieved clinically meaningful improvement in key osteoarthritis outcomes. If so, they remain at STEP 1. If not, they move on to STEP 2, which adds telephone-based coaching. Participants are assessed again three months later. Those that still have not achieved clinically relevant improvement move on to STEP 3, which adds a series of in-person physical therapy visits.
  Stepped Exercise Program: STEP 1: Participants have access to an internet-based exercise program for knee OA.
  STEP 2: Participants have access to an internet-based exercise program for knee OA plus telephone support.
  STEP 3: Participants have access to an internet-based exercise program for knee OA plus in-person physical therapy visit
- Arthritis Education (AE): The arthritis education intervention will include bi-weekly mailings of low-literacy educational materials on a comprehensive set of topics related to osteoarthritis and its management, based on established treatment guidelines.
Period: 3-Month Follow-Up
Arm/Group | STEP-KOA | Arthritis Education (AE)
Started | 230 | 115
Completed | 164 | 100
Not Completed | 66 | 15
Period: 6-Month Follow-Up
Arm/Group | STEP-KOA | Arthritis Education (AE)
Started | 209 (21 participants withdrew/excluded by 3-months, others missed that assessment but remained in study) | 113 (2 participants withdrew/excluded by 3-months, others missed that assessment but remained in study)
Completed | 164 | 100
Not Completed | 45 | 13
Period: 9-Month Follow-Up (Primary)
Arm/Group | STEP-KOA | Arthritis Education (AE)
Started | 196 (34 withdrew/excluded before 9 months; others missed prior assessments but remained in study) | 111 (4 withdrew/excluded before 9 months; others missed prior assessments but remained in study)
Completed | 163 (13 withdrew/refused before 9 months; others missed prior assessments but remained in study) | 95
Not Completed | 33 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STEP-KOA | Arthritis Education (AE) | Total
Number analyzed (Participants) | 230 | 115 | 345
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.9 (9.9) | 60.2 (11.1) | 60.0 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 15 | 45
  Male | 200 | 100 | 300
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 4 | 8
  Not Hispanic or Latino | 224 | 109 | 333
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 142 | 66 | 208
  White | 72 | 39 | 111
  More than one race | 11 | 6 | 17
  Unknown or Not Reported | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC)
Description: This is a measure of lower extremity pain (5 items), stiffness (2 items), and function (17 items), with items rated on a Likert scale of 0 (no symptoms) to 4 (extreme symptoms). The total scale range is 0-96, and higher scores mean a worse outcome.
Time Frame: Change from baseline to 3-month, 6-month, 9-month follow-ups. For STEP-KOA only, change from 9-month to 15-month follow-up.
Population: Intent to treat. Only the STEP-KOA group was assessed at 15 months. This was planned because the AE group could start receiving treatment after 9 months.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | STEP-KOA | Arthritis Education (AE)
Number analyzed (Participants) | 230 | 115
units on a scale
  Mean Change Scores from Baseline to 3-months | -4.85 (1.00) | 0.26 (1.27)
  Mean changes scores from baseline to 6-months | -3.97 (1.20) | -2.53 (1.54)
  Mean change scores from baseline to 9-months | -5.46 (1.15) | 1.38 (1.49)
  Mean change scores from 9 months to 15-months: number analyzed (Participants) | 230 | 0
  Mean change scores from 9 months to 15-months | 3.02 (1.38) |
Statistical Analysis 1: Comparison: STEP-KOA vs Arthritis Education (AE); This analysis of between-group difference in change from baseline to 3-month follow-up. We have not included a p-value because there was no pre-specified hypothesis for this time point. Rather, these are additional data obtained from the overall model, for which the 9-month time point was primary and included a pre-specified hypothesis; Test type: Other — As noted above, a statistical test was not specified at this time point. Rather, the data for all time points were included in the model and are presented here descriptively; Mean Difference (Final Values) = -5.1, 95% CI 2-sided [-8.2 to -2.0]
Statistical Analysis 2: Comparison: STEP-KOA vs Arthritis Education (AE); This is the analysis of between-group difference in change from baseline to 6-month follow-up. We have not included a p-value because there was no pre-specified hypothesis for this time point. Rather, these are additional data obtained from the overall model, for which the 9-month time point was primary and included a pre-specified hypothesis; Test type: Other — [test comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.4, 95% CI 2-sided [-5.2 to 2.3]
Statistical Analysis 3: Comparison: STEP-KOA vs Arthritis Education (AE); This is the analysis of between-group difference in change from baseline to 9-month follow-up. This is the primary outcome assessment time point; Test type: Superiority; p = 0.0003, Mixed Models Analysis; Mean Difference (Final Values) = -6.8, 95% CI 2-sided [-10.5 to -3.2]

2. Secondary Outcome: 30-second Chair Stand
Description: The 30 second stair stand asks participants to rise and sit back down in a chair as many times as they can during that time period, without using hands or arms for support. Higher scores mean better outcome (e.g. more stands in 30 seconds).
Time Frame: Change from baseline to 9-month follow-up
Population: Intent to treat
Measure: Mean (Standard Error); unit: Number of chair stands
Arm/Group | STEP-KOA | Arthritis Education (AE)
Number analyzed (Participants) | 230 | 115
Number of chair stands | -0.23 (0.29) | -0.59 (0.37)
Statistical Analysis 1: Comparison: STEP-KOA vs Arthritis Education (AE); This is the analysis between-group difference in change from baseline to 9-month follow-up for the 30 second chair stand; Test type: Superiority; p = 0.43, Mixed Models Analysis; Mean Difference (Final Values) = 0.4, 95% CI 2-sided [-0.6 to 1.3]

3. Secondary Outcome: 40m Fast-paced Walk
Description: The 40m fast-paced walk is a timed test of walking twice back and forth (as fast as participants are able) over a 10m distance. Lower scores mean better outcome (e.g. faster walking speed).
Time Frame: Change from baseline to 9-month follow-up
Population: Intent to treat
Measure: Mean (Standard Error); unit: seconds
Arm/Group | STEP-KOA | Arthritis Education (AE)
Number analyzed (Participants) | 230 | 115
seconds | -0.72 (1.26) | 1.61 (1.57)
Statistical Analysis 1: Comparison: STEP-KOA vs Arthritis Education (AE); Test type: Other; p = 0.23, Mixed Models Analysis; Mean Difference (Final Values) = -2.3, 95% CI 2-sided [-6.1 to 1.5]

ADVERSE EVENTS:
Time Frame: 15 months for each participant
Description: Adverse events were typically identified when participants told a study team member, during a routine contact (e.g., intervention contact, follow-up assessment contact) that a health event occurred.
Arm/Group | STEP-KOA | Arthritis Education (AE)
All-Cause Mortality (participants affected / at risk) | 1/230 | 0/115
Serious Adverse Events (participants affected / at risk) | 23/230 | 7/115
Other Adverse Events (participants affected / at risk) | 3/230 | 0/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEP-KOA (N=230) | Arthritis Education (AE) (N=115)
Hospitalization due bypass of peripheral artery (Vascular disorders) | 1 (2) | 0 (0)
Hospitalization for lymphatic leak following peripheral artery bypass (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hospitzalization for cardiac stents (Cardiac disorders) | 0 (0) | 1 (1)
Fall leading to injury (not study related) (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Blood clot in leg (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heart block (Cardiac disorders) | 1 (1) | 0 (0)
Hernia surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hospitalization following car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emergency Department Visit due to twisted ankle (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Emergncy room visit due to swollen legs and chest pain (Cardiac disorders) | 1 (1) | 0 (0)
Adverse drug reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Persistent soreness following car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalziation due to flu symptoms (Infections and infestations) | 1 (1) | 0 (0)
Emergency room visit due to a cold (Infections and infestations) | 0 (0) | 1 (1)
Hospitalization due to infection after liver biopsy (Infections and infestations) | 1 (2) | 0 (0)
Prostate cancer diagnosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Emergency department visit for knee pain after falling out of bed (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Torn ligament in knee (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Mini-strokes (Nervous system disorders) | 1 (1) | 0 (0)
Emergency department visit for heat stroke (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Hospitalization for cardiac catheterization and complidcations (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization due to depression (Psychiatric disorders) | 0 (0) | 1 (1)
Hospital visit due to high blood pressure (Cardiac disorders) | 0 (0) | 1 (1)
Hospitalization due to aneurysm (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization due to vertigo (Nervous system disorders) | 1 (1) | 0 (0)
Emergency department visit due to atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Knee replacement surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STEP-KOA (N=230) | Arthritis Education (AE) (N=115)
Fall with minor injuries (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Increased hip pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-03-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02653768/Prot_SAP_001.pdf
  • Informed Consent Form (2016-10-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT02653768/ICF_000.pdf